CLINICAL TRIAL: NCT00355225
Title: Community-Effectiveness of the Distribution of Insecticide-Treated Bed Nets Through Social Marketing Antenatal Care Services in Malaria Control in Rural Burkina Faso
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: SFB544D4
Record Dates: First submitted 2006-07-19; First posted 2006-07-21 (Estimated); Last update posted 2006-10-09 (Estimated); Status verified 2006-07

CONDITIONS: Malaria
Keywords: insecticide-treated bednets; malaria; africa; social marketing; ante-natal care; ITN coverage; ITn use
MeSH Terms: conditions — Malaria

INTERVENTIONS:
Procedure: ITN distribution channel

SUMMARY:
The study aims at assessing which of two distribution channels for insecticide treated bendnets (ITNs), social marketing vs. social marketing coupled with free distribution through ante-natal care, is most effective in reaching groups at high risk of malaria, i.e. pregnant women and children under 5.

DETAILED DESCRIPTION:
The hypothesis that insecticide-treated bed net (ITN) effects may not be long-lasting in young children living in areas of intense malaria transmission due to interactions with the immunologi-cal development has now been refuted in a number of studies including the D4 study. The highly controversial question remains how African programmes can best reach a sustainable high coverage with ITNs in young children and pregnant women. Against this background it is planned to implement a cluster randomised controlled trial in Nouna Health District in Burkina Faso. Twenty-two peripheral health centres and their catchment areas will be randomised to (1) ITN provision to the general population through social marketing and (2) ITN provision to the general population through social marketing plus free provision to all pregnant women through antenatal services. The primary outcomes are ITN coverage in households and ITN use during pregnancy and infancy.

ELIGIBILITY:
Inclusion Criteria:

* Being one of 25 primary health facility catchment areas in the Nouna Health District, Burkina Faso

Exclusion Criteria:

* Being outside one of 25 primary health facility catchment areas in the Nouna Health District, Burkina Faso

Min Age: 0 Years | Sex: All
Age Groups: Child, Adult, Older Adult

PRIMARY OUTCOMES:
ITN coverage in households 12 and 24 months after the start of the interventions
ITN use during pregnancy and infancy

SECONDARY OUTCOMES:
Costs per malaria case and per DALY prevented
Self-reported information on ANC visits
Insecticide content on ITN and mortality of vector mosquitoes over time
Acceptance of health staff and population

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Mueller, MD, MPH, Principal Investigator — Heidelberg University